CLINICAL TRIAL: NCT02560077
Title: Study the Effect of Cashew Apple Juice on the Physiological and Psychological Fitness in the Middle Aged and Elderly Volunteers
Brief Title: Effect of Cashew Apple Juice on the Physiological and Psychological Fitness in the Middle Aged and Elderly Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Jintanaporn Wattanathorn, Integrative complementary alternative medicine, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: HE 531319
Record Dates: First submitted 2015-04-11; First posted 2015-09-25 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
Keywords: cognitive; memory; physical fitness; psychological fitness; elderly; middle aged

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- placebo (Placebo Comparator): The placebo and cashew apple fruit juice had the same color and smell
  Interventions: Other: placebo
- cashew apple juice 120 mg/day (Active Comparator): The subjects who were assigned as the low dose treatment group received cashew apple fruit juice extract at dose of 120 mg/day
  Interventions: Other: cashew apple juice
- cashew apple juice 240 mg/day (Active Comparator): The subjects who were assigned as the high dose treatment group received cashew apple fruit juice extract at dose of 240 mg/day
  Interventions: Other: cashew apple juice

INTERVENTIONS:
Other: placebo — Subject receive the Placebo product (placebo group had same color and smell of treatment groups)
  Arms: placebo
Other: cashew apple juice — Subject received the cashew apple juice at dose of 120 mg/day after meal
  Arms: cashew apple juice 120 mg/day
Other: cashew apple juice — Subject received the cashew apple juice at dose of 240 mg/day after meal
  Arms: cashew apple juice 240 mg/day

SUMMARY:
Cashew or Anacardium occidentale L. is a plant in a family of Anacardiaceae. The fruit of cashew or cashew apple may be consumed fresh, but contains high quantities of tannins yielding a bitter taste and dry mouth feel. Therefore, it is more often prepared as beverage. It is rich in carbohydrate and vitamin C. It is also claimed for numerous ailments including antitumor, antimicrobial, urease inhibitory and lipoxygenase activity. In addition, cashew apple juice also has excellent anti-oxidant potential. The preclinical data also demonstrated that cognitive deficit rats induced by cholinotoxin which received A.occidentale or cashew fruit juice for 2 weeks showed the neuroprotective and cognitive enhancing effects.Therefore, the potential benefit of Cashew apple juice on physical fitness and psychological fitness of the middle aged and elderly is focused.

DETAILED DESCRIPTION:
Currently, the age-related health problems are increasing their importance markedly due to the increased elderly population. These problems produce the great socio-economic burdens of country. In addition, the quality of both the elderly and their families are also decreased. Therefore, the anti-aging strategy for the elderly has gained much attention. Based on the role of oxidative stresses and free radicals on the age-related pathology, the development of anti-aging health products from substances possessing antioxidant effect has been focused.

Cashew or Anacardium occidentale Linn, one of the economic plants in Thailand, is originated from Latin America and possesses antioxidant effect. In Latin America, this plant is used as anti-aging and memory enhancer. Data obtained from animal study also showed that cashew apple juice could enhance memory and increased muscle performance and induced fatigue resistance. Therefore, cashew apple has the potential to be developed as the physical and psychological fitness enhancer heath product for the elderly. However, no scientific data are available until now. Therefore, this study aimed to develop the cashew apple juice based functional drink and to determine the effect of 12- week consumption of cashew apple juice on physical and psychological fitness of the middle aged and elderly volunteers. The consumption safety of the developed drink was also investigated.

The developed cashew apple juice based functional drink showed antioxidant and acetylcholinesterase suppression activities. Therefore, it was used for the investigation the effect of 12- week consumption of cashew apple juice on physical and psychological fitness of the middle aged and elderly volunteers. In this study, the healthy middle aged and elderly volunteers who were recruited to participate in this study were divided in to various groups consisting of placebo and the Cashew drink treated groups at doses of 120 and 240 mg/day. All subjects had to consume the assigned drinks for 12 weeks. They were determined the parameters related to physical and psychological fitness before treatment and every 4 weeks throughout the study period. The assessments were also performed at 4 week after the cessation of cashew apple juice based drink consumption. The physical fitness assessment was performed via the battery test consisting of various tests including 30-second chair stand test which measured the muscle strength of the lower extremities, hand grip strength test which measured the muscle strength of hand, 6-minute walk test which measured cardio-pulmonary endurance and Tandem test which measured postural balance. The alteration of oxidative stress markers including the malondialdehyde level and the activities of superoxide dismutase (SOD), catalase (CAT) and glutathione peroxidase (GSH-Px) in blood was also motored. The results showed that the volunteers who consumed cashew apple juice based drink at dose of 240 mg/day improved the performance in 30-second chair stand test and 6-minute walk test at 12 weeks of consumption period. The enhanced GSH-Px activity and the decreased MDA level were also observed. Therefore, the data obtained from this study demonstrated the increased muscle strength of the lower extremities and the cardio-pulmonary endurance of the middle-aged and elderly volunteers. The possible underlying mechanism might occur partly via the improved oxidative stress status.

In order to evaluate the psychological fitness, the working memory was assessed using computerized battery test while the attention and cognitive processing were assessed via event related potential. Emotion was assessed via Bond-Läder test whereas psychological symptoms were evaluated by symptoms checklist-90 (SCL-90). In addition, the functions of cholinergic and monoaminergic system especially dopamine were also evaluated using the activities of acetylcholinesterase (AChE), monoamine oxidase (MAO B) as indices respectively. The assessments were performed at the same time schedules as the physical assessment. The results showed that the subjects who consumed cashew apple juice based drink at dose of 240 mg/day showed the following changes; 1) working memory was improves in all domains including the increased power of attention, the increase continuity of attention, the speed of memory and the quality of memory 2) the decreased latency but increased amplitude of N100 and P300 3) the suppression of AChE and MAO-B. Therefore, the current data revealed that the volunteers who consumed the cashew apple juice based drink at dose of 240 mg/day enhance attention and cognitive processing ability giving rise to the improved working memory. The possible underlying mechanism might occur partly via the improved cholinergic and dopaminergic functions.

When the quality of life was determined by using Quest quality questionnaire which modified from SF-36 at the end of study, the results showed that volunteers who consumed cashew apple juice based drink showed the higher quality of life than the volunteer who consumed placebo. These suggested that the cashew apple juice based drink improved both physical and psychological fitness and quality of life of the middle-aged and elderly volunteers.

In order to assure the consumption safety of the consumers, the assessments of hematological and chemical changes of the volunteers were also performed. The results showed that no toxicity was observed throughout the study period. The results obtained from this study demonstrated that the cashew apple juice based drink improved physical and psychological fitness together with the quality of life without toxicity. Therefore, the developed cashew apple juice based drink has the potential to be served as the functional drink in order to enhance physical and psychological fitness for the middle-aged and elderly.

ELIGIBILITY:
Inclusion Criteria:

* Live in Khon Kaen, Thailand
* Aged between 55-70 years old
* Body mass index is 18.5 to 24.9
* Signed a written consent form
* In order to ensure the healthy condition , all subjects were subjected to history interviewed by the semi structure form. Moreover they all were assessed physical exam by physician
* All volunteers should not use other nutraceutical compounds or herbs or drugs which influenced on the nervous system function at least 1 month before participating in this study
* On the day of the study, all volunteers felt well and refrain from drinking tea or coffee, or smoking more than 10 pieces/ day

Exclusion Criteria:

* Cardiovascular disease
* Respiratory disease
* Neuropsychological disorders
* Diabetes
* Liver disease
* Renal disease
* Endocrine dysfunction
* Autoimmune disease
* Hematological disorder
* Cancer
* Brain inflammation, head injury

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-12; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Cognitive processing (P300) and attention (N100) using Event Related Potential | 4 months

SECONDARY OUTCOMES:
Accuracy and speed of working memory using computerized battery test | 4 months
Mood evaluation using Bond-laddeer questionnaire | 4 months
Psychological symptom using SCL-90 questionnaire | 4 months
Malondialdehyde level (MDA) in the serum | 4 months
Acetylcholinesterase and monoamine oxidase-B activities in serum | 4 months
Superoxide dismutase (SOD), catalase (CAT), glutathione peroxidase activity (GSH-Px) in the serum | 4 months
Strength of lower extremities muscles using 30 second chair stand test | 4 months
Upper body muscular strength using Hand grip strength test | 4 months
Cardio-pulmonary endurance using 6-minute walk test | 4 months
Static balance using Tandem stance test | 4 months
The changes of hematological and clinical chemistry parameters | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Jintanaporn Wattanathorn, Principal Investigator — Integrated complementary alternative medicine